CLINICAL TRIAL: NCT00169039
Title: Clozapine Response and Biogenic Amines in Schizophrenia
Brief Title: Clozapine Versus Chlorpromazine for Treatment-Unresponsive Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Dartmouth-Hitchcock Medical Center (Other); Commonwealth Research Center, Massachusetts (Other); Novartis (Industry)
Responsible Party: Principal Investigator, AlanGreen, Chair, Department of Psychiatry Geisel School of Medicine at Dartmouth, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH049891 (NIH); R01MH049891 (NIH)
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
Keywords: Clozapine; Chlorpromazine; Schizophrenia; Biochemistry
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine; Chlorpromazine

INTERVENTIONS:
Drug: Clozapine
Drug: Chlorpromazine

SUMMARY:
This study will examine the physical response to clozapine or chlorpromazine in people with schizophrenia that has not improved with treatment.

DETAILED DESCRIPTION:
This is a longitudinal double-blind 12-week study of the clinical and biochemical response to clozapine or chlorpromazine in a group of treatment-refractory schizophrenic patients.

The study has 4 phases: (1) A recruitment period; (2) a period of discontinuation of psychotropic medication; (3) a drug-washout period; and (4) a 12-week double-blind trial of clozapine or chlorpromazine.

ELIGIBILITY:
Inclusion Criteria:

* 19-60 years of age
* Diagnosis of schizophrenia
* BPRS score > 50
* Clinical Global Impressions rating > 4
* One of the following: BPRS items rated greater than or equal to 4, conceptual disorganization, suspiciousness, hallucinations, unusual thought content.
* At least 2 six-week trials of different neuroleptics given at a dosage equivalent to at least 600 mg per day of chlorpromazine OR at least 1 eight-week trial of a neuroleptic given at a dosage equivalent to at least 800 mg per day of chlorpromazine.
* The patient (or the patient's authorized legal representative) must understand the nature of the study and sign the informed consent.

Exclusion Criteria:

* History of substance dependence within the past 2 months
* Major medical problems precluding the use of clozapine
* Pregnancy or lactation
* A serious suicide/homicide risk

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66
Dates: Start 1994-12; Study Completion 2002-02

PRIMARY OUTCOMES:
Clinical measures: Brief Psychiatric Rating Scale, Clinical Global Impression, Scale for the Assessment of Negative Symptoms, Simpson-Angus Scale, Abnormal Involuntary Movement Scale and Barnes Akathisia Scale.

SECONDARY OUTCOMES:
Biological measures: plasma and urinary samples of dopamine, norepinephrine and their metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Alan I Green, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Commonwealth Research Center, Jamaica Plain, Massachusetts, United States

REFERENCES:
- [Background] Green AI, Alam MY, Boshes RA, Waternaux C, Pappalardo KM, Fitzgibbon ME, Tsuang MT, Schildkraut JJ. Haloperidol response and plasma catecholamines and their metabolites. Schizophr Res. 1993 Jun;10(1):33-7. doi: 10.1016/0920-9964(93)90074-s. PMID 8369230
- [Background] Green AI, Alam MY, Sobieraj JT, Pappalardo KM, Waternaux C, Salzman C, Schatzberg AF, Schildkraut JJ. Clozapine response and plasma catecholamines and their metabolites. Psychiatry Res. 1993 Feb;46(2):139-49. doi: 10.1016/0165-1781(93)90016-a. PMID 8483973